CLINICAL TRIAL: NCT00664521
Title: A Randomized, Double-blind, Placebo Controlled, Multi-centre, Exploratory, Pilot, Phase II Trial of 150mg Atacicept Given Subcutaneously in Combination With Rituximab in Subjects With Rheumatoid Arthritis.
Brief Title: Atacicept in Combination With Rituximab in Subjects With Rheumatoid Arthritis (August III)
Acronym: August III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28155
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rituximab Plus Atacicept (Experimental): Rituximab will be administered as an intravenous infusion at a dose of 1000 mg at Weeks 1 and 3, followed by atacicept 150 mg subcutaneously once a week from Week 7 to 32.
  Interventions: Biological: Rituximab; Drug: Atacicept
- Rituximab Plus Placebo (Placebo Comparator): Rituximab will be administered as an intravenous infusion at a dose of 1000 mg at Weeks 1 and 3, followed by placebo matched to atacicept subcutaneously once a week from Week 7 to 32.
  Interventions: Biological: Rituximab; Drug: Placebo matched to atacicept

INTERVENTIONS:
Biological: Rituximab — Rituximab will be administered as an intravenous infusion at a dose of 1000 mg at Weeks 1 and 3.
Drug: Atacicept — Atacicept will be administered at a dose of 150 mg subcutaneously once a week from Week 7 to 32.
  Arms: Rituximab Plus Atacicept
Drug: Placebo matched to atacicept — Placebo matched to atacicept will be administered subcutaneously once a week from Week 7 to 32.
  Arms: Rituximab Plus Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of combined treatment with atacicept and rituximab in subjects with active rheumatoid arthritis (RA) receiving re-treatment with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Greater than and equal to (>=) 18 years of age at the time of Informed Consent
* Who have rheumatoid arthritis satisfying American College of Rheumatology (ACR) criteria with a disease history of at least 12 months
* Subjects must have active disease defined by DAS28 >3.2
* Subjects must have received previous treatment with rituximab and must be candidates for re-treatment with rituximab
* Female subjects of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for 4 weeks before study day 1 (SD1), during the treatment period and for 12 months after the last dose of rituximab, and must have a negative urine pregnancy test at the screening visit and SD1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Current neurological disease excluding migraine
* Inflammatory joint disease other than rheumatoid arthritis
* Any contraindication to rituximab as per national label
* Use of disease-modifying anti-rheumatic drugs (DMARDs; including methotrexate) for less than 3 months or change in dosing regimen within 28 days before SD1, or methotrexate dose regimen >25 mg/week
* Participation in any interventional clinical trial within 1 month before SD1 (or within 5 half-lives of the investigated compound before SD1, whichever is longer)
* Prednisone dose regimen >10 mg/day (or equivalent), or change in steroid dosing regimen within 28 days before SD1
* Active or latent tuberculosis within the year before screening or major infection requiring hospitalization or intravenous anti-infectives within 28 days before SD1
* Serum Immunoglobulin G (IgG) below 6 gram per liter (g/L)
* Known hypersensitivity to atacicept or to any of the components of the formulated atacicpet
* Known hypersensitivity to rituximab, to any of the components of the formulated rituximab or to murine proteins
* Breastfeeding or pregnancy
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- France (3):
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Strasbourg
- Research Site, Amsterdam, Netherlands
- Sweden (2):
  - Research Site, Malmo
  - Research Site, Stockholm
- United Kingdom (2):
  - Research Site, Newcastle
  - Research Site, Norwich

REFERENCES:
- [Result] van Vollenhoven RF, Wax S, Li Y, Tak PP. Safety and efficacy of atacicept in combination with rituximab for reducing the signs and symptoms of rheumatoid arthritis: a phase II, randomized, double-blind, placebo-controlled pilot trial. Arthritis Rheumatol. 2015 Nov;67(11):2828-36. doi: 10.1002/art.39262. PMID 26137975

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus Atacicept: Rituximab was administered as an intravenous infusion at a dose of 1000 milligram (mg) at Weeks 1 and 3, followed by atacicept 150 mg subcutaneously once a week from Week 7 to 32.
- Rituximab Plus Placebo: Rituximab was administered as an intravenous infusion at a dose of 1000 milligram (mg) at Weeks 1 and 3, followed by placebo matched to atacicept subcutaneously once a week from Week 7 to 32.
Period: Overall Study
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Started | 18 | 9
Completed | 12 | 8
Not Completed | 6 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.0) | 57.7 (11.5) | 57.2 (11.0)
Gender [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Baseline up to Week 64
Population: Safety population included all participants who received at least one dose of atacicept or placebo.
Measure: Number; unit: Participants
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 18 | 9
Participants
  AEs | 17 | 9
  SAEs | 6 | 2

2. Primary Outcome: Percentage of Participants With Immunoglobulin G (IgG) Level Less Than 3 Gram Per Liter (g/L)
Time Frame: Week 64
Population: Safety population included all participants who received at least one dose of atacicept or placebo. Here. "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 11 | 5
percentage of participants | 0 | 0

3. Primary Outcome: Percent Change From Baseline in Vital Signs and Routine Safety Lab Parameters at Week 32
Description: Vital signs assessed included blood pressure (systolic and diastolic), pulse and body temperature. Routine safety lab parameters evaluated included red blood cell (RBC), hemoglobin, hematocrit, platelets, mean cellular hemoglobin (MCH), MCH concentration, MCH volume, white blood cell (WBC), lymphocytes, monocytes, eosinophils, basophils, neutrophils, gamma glutamyl transferase (GGT), alanine aminotransferase (ALT), albumin, alkaline phosphatase (AP), aspartate aminotransferase (AST), bilirubin, calcium, creatinine, glucose, potassium, total protein, sodium, uric acid, and blood urea nitrogen. Percent change from baseline was calculated as ([Week 32 value minus baseline value] multiplied by 100) divided by baseline value.
Time Frame: Baseline, Week 32
Population: Safety population included all participants who received at least one dose of atacicept or placebo. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 12 | 9
Percent change
  Systolic Blood Pressure (n = 12, 9) | 3.74 (11.76) | -6.29 (13.80)
  Diastolic Blood Pressure (n = 12, 9) | 1.09 (11.19) | 4.89 (10.09)
  Pulse (n = 12, 9) | 10.21 (19.93) | -8.54 (11.98)
  Temperature (n = 10, 8) | 0.23 (1.05) | -0.44 (0.86)
  RBC (n = 12, 9) | 3.10 (5.30) | 4.94 (7.18)
  Hemoglobin (n = 12, 9) | 2.55 (5.32) | 4.93 (6.18)
  Hematocrit (n = 12, 9) | 2.39 (6.30) | 6.05 (6.15)
  Platelets (n = 12, 9) | -6.80 (21.21) | -2.49 (37.62)
  MCH (n = 12, 9) | -0.32 (5.03) | 0.22 (3.21)
  MCH Concentration (n = 12, 9) | -0.18 (2.01) | -1.41 (1.47)
  MCH Volume (n = 12, 9) | -0.06 (4.98) | 1.39 (2.73)
  WBC(n = 12, 9) | -14.59 (36.85) | -9.70 (19.15)
  Lymphocytes (n = 12, 9) | 0.27 (30.11) | -5.68 (23.00)
  Monocytes (n = 12, 9) | 5.01 (70.44) | 1.88 (38.51)
  Eosinophils (n = 12, 9) | 34.11 (103.78) | -7.51 (34.58)
  Basophils (n = 12, 9) | -20.45 (58.61) | 32.41 (117.44)
  Neutrophils (n = 12, 9) | -11.29 (57.75) | -13.09 (24.01)
  GGT (n = 12, 9) | -3.21 (30.37) | 10.17 (53.33)
  ALT (n = 12, 9) | 17.52 (27.89) | 17.79 (53.23)
  Albumin (n = 12, 9) | 6.22 (6.34) | 6.43 (8.10)
  AP (n = 12, 9) | 4.85 (18.86) | -5.41 (16.48)
  AST (n = 12, 9) | 14.53 (30.87) | 6.73 (36.47)
  Bilirubin Total (n = 12, 9) | 15.09 (42.78) | 4.76 (14.29)
  Calcium (n = 12, 9) | -1.07 (5.04) | 2.61 (4.72)
  Creatinine (n = 12, 9) | -3.29 (10.30) | 5.89 (5.26)
  Glucose (n = 12, 9) | 3.71 (18.55) | 7.99 (22.71)
  Potassium (n = 12, 9) | -0.93 (6.34) | 4.67 (9.37)
  Total Protein (n = 12, 9) | -2.83 (7.08) | 4.17 (6.57)
  Sodium (n = 12, 9) | 1.21 (1.46) | 0.25 (1.63)
  Uric Acid (n = 12, 9) | -2.95 (12.60) | -0.72 (6.10)
  Blood Urea Nitrogen (n = 12, 9) | 1.63 (27.04) | -7.42 (26.02)

4. Primary Outcome: Percent Change From Baseline in Anti-tetanus and Anti-diphteria Immunization Titer at Week 32
Description: Percent change from baseline was calculated as ([Week 32 value minus baseline value] multiplied by 100) divided by baseline value.
Time Frame: Baseline, Week 32
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 10 | 9
percent change
  Anti-tetanus Immunization Titer | -17.98 [-34.29 to 0.00] | 0.00 [-7.67 to 23.68]
  Anti-diphtheria Immunization Titer | -33.68 [-50.00 to 0.00] | 8.41 [0.39 to 33.93]

5. Primary Outcome: Percent Change From Baseline in Anti-pneumococcus Titer at Week 32
Description: as for outcome 4
Time Frame: Baseline, Week 32
Population: Safety population included all participants who received at least one dose of atacicept or placebo. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 10 | 9
percent change | -18.49 [-35.18 to 0.00] | 0.00 [0.00 to 0.00]

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Response Based on C-reactive Protein (ACR20-CRP), ACR50-CRP and ACR70-CRP at Week 32
Description: ACR20-CRP response: greater than or equal to (>=) 20 percent (%) improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=20% improvement in at least 3 of the following: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP). ACR50-CRP and ACR70-CRP response are defined as >=50% and >=70% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) respectively together with >=50% and >=70% improvement in at least 3 of the following respectively: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) CRP.
Time Frame: Week 32
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 18 | 9
percentage of participants
  ACR20-CRP | 33.3 | 22.2
  ACR50-CRP | 11.1 | 11.1
  ACR70-CRP | 5.6 | 0

7. Secondary Outcome: Change From Baseline in Disease Activity Score in 28 Joints (DAS28) Based on CRP (DAS28-CRP) at Week 32
Description: DAS28-CRP incorporates non-graded joint counts for tenderness and swelling based on a total of 28 joints, CRP as a marker of inflammation, and a general health assessment using a 100 mm visual analog scale (the participant's global assessment of disease activity). DAS28 score ranges between 0 and 10 representing current disease activity. A value above 5.1 represents high disease activity, a value below 3.2 represents low disease activity, and a value below 2.6 represents remission.
Time Frame: Baseline, Week 32
Population: ITT population included all randomized participants. Here 'n' signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 18 | 9
Units on a scale
  Baseline (n = 18, 9) | 5.50 (0.99) | 5.81 (1.04)
  Change at Week 32 (n = 12, 9) | 3.85 (0.98) | 4.25 (1.10)

8. Secondary Outcome: Median Percentage Change From Baseline in Levels of Total, Mature and Memory B Cells
Description: Flow cytometric analysis of lymphocyte populations using four-color fluorescence-activated cell sorting was performed for the analysis of total, mature and memory B cell levels.
Time Frame: Baseline, Week 3, 7, 12, 16, 26 and 32
Population: Safety population included all participants who received at least one dose of atacicept or placebo. Here 'n' signifies those participants who were evaluable for the specified category.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Number analyzed (Participants) | 18 | 9
percent change
  Total B cells (Week 3: n=18, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Total B cells (Week 7: n=17, 8) | -100.00 [-100.00 to -100.00] | -99.69 [-100.00 to -96.96]
  Total B cells (Week 12: n=16, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Total B cells (Week 16: n=15, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Total B cells (Week 26: n=12, 9) | -100.00 [-100.00 to -93.06] | -94.74 [-100.00 to -71.43]
  Total B cells (Week 32: n=12, 9) | -86.99 [-98.26 to -50.00] | -68.11 [-100.00 to -35.00]
  Mature B Cells (Week 3: n=18, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Mature B Cells (Week 7: n=17, 8) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Mature B Cells (Week 12: n=16, 9) | -100.00 [-100.00 to -47.78] | -100.00 [-100.00 to -100.00]
  Mature B Cells (Week 16: n=15, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Mature B Cells (Week 26: n=12, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -85.11]
  Mature B Cells (Week 32: n=12, 9) | -99.35 [-100.00 to -22.73] | -84.47 [-100.00 to -48.94]
  Memory B cells (Week 3: n=18, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Memory B cells (Week 7: n=17, 8) | -100.00 [-100.00 to -66.67] | -100.00 [-100.00 to -100.00]
  Memory B cells (Week 12: n=16, 9) | -100.00 [-100.00 to -68.33] | -100.00 [-100.00 to -100.00]
  Memory B cells (Week 16: n=15, 9) | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -66.67]
  Memory B cells (Week 26: n=12, 9) | -100.00 [-100.00 to -82.50] | -88.89 [-100.00 to -25.00]
  Memory B cells (Week 32: n=12, 9) | -83.33 [-100.00 to -25.00] | -50.00 [-100.00 to -44.44]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 64
Arm/Group | Rituximab Plus Atacicept | Rituximab Plus Placebo
Serious Adverse Events (participants affected / at risk) | 6/18 | 2/9
Other Adverse Events (participants affected / at risk) | 17/18 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus Atacicept (N=18) | Rituximab Plus Placebo (N=9)
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Demyelination (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint capsule rupture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus Atacicept (N=18) | Rituximab Plus Placebo (N=9)
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Influenza (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Injection site reaction (General disorders) | 7 | 2
Injection site erythema (General disorders) | 4 | 0
Injection site pruritus (General disorders) | 4 | 0
Injection site swelling (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Injection site pain (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Injection site irritation (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Type I hypersensitivity (Immune system disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Weight increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results, Institution and Principal Investigator (PI) must first provide Sponsor with a copy of proposed publication for review at least 30 days prior to submission. If Institution and PI do not agree to modification, they shall so notify Sponsor and postpone submission for additional 60 days to allow Sponsor to seek legal remedies or file patent applications. There is a need for coordinated approach to any publication of results from sites for any multi-site study.